CLINICAL TRIAL: NCT01748162
Title: Management of Recurrent Croup: Comparison Between Inhaled Fluticasone and Oral Prednisolone
Brief Title: Management of Recurrent Croup
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, David Brown, Associate Professor of Otorhinolaryngology, University of Michigan
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 00059385
Record Dates: First submitted 2012-10-31; First posted 2012-12-12 (Estimated); Results first posted 2017-11-13 (Actual); Last update posted 2017-11-13 (Actual); Status verified 2017-11

CONDITIONS: Croup
Keywords: croup; recurrent croup; barky cough
MeSH Terms: conditions — Croup | interventions — Fluticasone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Inhaled steroids (Experimental): Daily inhaled steroids. Fluticasone 2 puffs inhaled orally twice daily for six months.
  Interventions: Drug: Fluticasone
- Oral control (Active Comparator): Patient and clinician observation with short term oral prednisolone as needed. Offered at 1mg/kg (body weight) daily dosing for symptomatic treatment on as needed basis for three days, but may be modified per managing physician's discretion.
  Interventions: Drug: Prednisolone IF needed

INTERVENTIONS:
Drug: Fluticasone — Daily inhaled steroids. Fluticasone 2 puffs inhaled orally twice daily for six months.
  Arms: Inhaled steroids
Drug: Prednisolone IF needed
  Arms: Oral control

SUMMARY:
Presently children who experience recurring croup symptoms receive a variety of treatments. This is because it is not clear which treatments may be best. Some children are given inhaled steroids (similar to what children with asthma use). Others are carefully watched and cautioned to avoid potential triggers (certain foods, environmental allergens, etc), and should episodes of croup recur they are treated with a short course of oral steroids. The purpose of this study is to compare two safe and clinically appropriate methods for treating recurrent croup, daily inhaled steroids versus observation with oral steroids on an as needed basis, to see if either is useful in preventing future episodes of croup.

ELIGIBILITY:
Inclusion Criteria:

* Pediatric population: 6 months to 15 years of age
* 2 or more episodes of croup in 12 month period

  * croup defined as acute onset inspiratory stridor, barking cough, with respiratory distress.

Exclusion Criteria:

* Grade 3 or 4 subglottic stenosis
* Subglottic hemangioma
* Posterior laryngeal cleft
* Recurrent respiratory papillomatosis
* External compression (Innominate artery compression, mediastinal mass, (double aortic arch, etc)
* Symptoms or signs suggesting another cause of stridor, such as epiglottitis, bacterial tracheitis, or supraglottic foreign body
* Tracheomalacia/ bronchomalacia severe enough to cause respiratory distress
* Current steroid therapy for previously diagnosed condition, i.e. reactive airway disease.
* Other medical conditions necessitating chronic steroid utilization

Ages: 6 Months to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 10 (Actual)
Dates: Start 2012-09; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: David J Brown, MD, Principal Investigator — University of Michigan Department of Otolaryngology-Head & Neck Surgery
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

REFERENCES:
- See also: Please visit our Department Facebook page for information regarding the study — http://www.facebook.com/MichiganOtolaryngology

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 10 participants were recruited and consented and had their initial baseline bronchoscopy, but of the 5 at 1 site, only 1 had an actual croup episode within he first 6 months. Because of decreased recruitment, the study was terminated. The other site's data is not fully available due to unexpected staff turnover and systems failures.
Groups:
- Oral Control: Short term oral prednisolone. Offered at 1mg/kg daily dosing for symptomatic treatment on as needed basis for three days, but may be modified per managing physician's discretion.
Period: Overall Study
Arm/Group | Inhaled Steroids | Oral Control
Started | 5 | 5
Started 6 Month Initial Treatment Plan | 2 | 2
Completed 6 Month Initial Treatment | 0 | 0
Started 6 Month Followup | 0 (No participants in either arm had additional croup episodes in the first 6 months; study terminated.) | 0 (No participants in either arm had additional croup episodes in the first 6 months; study terminated.)
Completed | 0 | 0
Not Completed | 5 | 5
Not completed — no additional croup episodes to evaluate | 2 | 2
Not completed — participant consented but did not begin | 0 | 1
Not completed — reasons not available | 3 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Inhaled Steroids | Oral Control | Total
Number analyzed (Participants) | 5 | 5 | 10
Age, Customized [Count of Participants; unit: Participants] — Age brackets of children participating:
  Participants
    6 months to 15 years | 5 | 5 | 10
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Due to unexpected staff turnover, data from one site is incomplete.
  Participants
    number analyzed (Participants) | 2 | 3 | 5
    Female | 0 | 2 | 2
    Male | 2 | 1 | 3
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5 | 5 | 10

OUTCOME MEASURES:

1. Primary Outcome: Quantity of Recurrent Episodes
Description: Quantity of recurrent croup episodes experienced over a 1 year period by each participating subject.
Time Frame: 1 year
Population: No participants completed to 1 year because of early study termination.
Arm/Group | Inhaled Steroids | Oral Control
Number analyzed (Participants) | 0 | 0

2. Secondary Outcome: Severity of Croup Episodes
Description: Severity of recurrent croup episodes based on Westley Croup scale (0 - 17, where 0 is mildest croup symptoms and 17 is most severe symptoms.)
Time Frame: 1 year
Population: No participants completed to 1 year because of early study termination.
Arm/Group | Inhaled Steroids | Oral Control
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: Six months (because study was terminated based on no participants having additional episodes).
Arm/Group | Inhaled Steroids | Oral Control
Serious Adverse Events (participants affected / at risk) | 0/5 | 0/5
Other Adverse Events (participants affected / at risk) | 0/5 | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes